CLINICAL TRIAL: NCT00804323
Title: Semi-Automated Patterned Laser Trabeculoplasty
Brief Title: PASCAL Trabeculoplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APEC-041
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Open-Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Group 1 (Experimental): Patients with open-angle glaucoma
  Interventions: Procedure: Patter Scan Laser System (OptiMedica, Santa Clara, CA, USA)

INTERVENTIONS:
Procedure: Patter Scan Laser System (OptiMedica, Santa Clara, CA, USA) — Pattern Scan Laser trabeculoplasty

SUMMARY:
Argon laser trabeculoplasty (ALT) with 100 ms pulses is an effective therapy for lowering intraocular pressure (IOP). Similar reductions in IOP have been achieved using ns (SLT) and microsecond (MLT) pulses, which produce less thermal damage to trabecular meshwork (TM). Lack of clinically visible changes may make the accurate alignment of subsequent pulses difficult. We describe a novel technique - Patterned Laser Trabeculoplasty (PLT) using the PASCAL Photocoagulator system, and its preliminary evaluation in patients with open angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* 18-year-old patients
* Uncontrolled Open angle (Shaffer IV)
* No previous surgical trabeculoplasty or glaucoma surgery

Exclusion Criteria:

* Patients not willing to participate
* Angle-closure glaucoma
* No clear optical media

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-12 (Actual); Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Intraocular Pressure | During follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Felix Gil Carrasco, MD, Principal Investigator — Asociación para Evitar la Ceguera en México
Locations (1):
- Asociación para Evitar la Ceguera en México, Mexico City, Mexico City, Mexico